CLINICAL TRIAL: NCT07257978
Title: A Phase II/III Double-blind, Randomised, Placebo-controlled, Crossover Study Investigating the Efficacy and Safety of NTI164 in Children and Young Adults With Rett Syndrome
Brief Title: Efficacy and Safety of NTI164 in Children and Young Adults With Rett Syndrome
Acronym: TRANSCEND
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fenix Innovation Group (Industry)
Collaborators: Neurotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTIRTT2; NTIRTT2 (Other: Fenix Innovation Group Pty Ltd)
Record Dates: First submitted 2025-07-18; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: RETT Syndrome With Proven MECP2 Mutation; Rett Syndrome
Keywords: Rett syndrome; Rett; cannabis; NTI164
MeSH Terms: conditions — Rett Syndrome; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled, double-blind, crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties other than the Clinical Trials Pharmacy and Sponsor will be blinded during the Active study phase (up to Week 28).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- NTI164 active (Active Comparator): NTI164
  Interventions: Drug: NTI164

INTERVENTIONS:
Drug: NTI164 — NTI164 is a full-spectrum medicinal cannabis plant extract with <0.3% THC.
  Other Names: FEN164
  Arms: NTI164 active
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The FENRTT2 study will investigate the efficacy and safety of a medicinal cannabis plant extract with extremely low THC (delta-9-tetrahydrocannabinol), NTI164, on Rett syndrome (RTT) in a crossover design. RTT is a devastating rare genetic condition affecting females and involves debilitating physical and intellectual symptoms. NTI164 is an oil which has demonstrated efficacy in reducing symptoms in several paediatric neurological conditions, including RTT, autism spectrum disorder (ASD), and paediatric acute-onset neuropsychicatric syndrome (PANS). A Phase I/II clinical trial of NTI164 in RTT (FENRTT1/NTIRTT1) showed NTI164 is safe in this population and significantly improved overall clinical severity of illness, as well as core RTT symptoms, including anxiety, mental alertness, communication skills, socialisation/eye contact, and attentiveness. The FENRTT2 study will investigate NTI164 in a larger number of patients, and compare NTI164 to a placebo control. Research tests on patient blood will also be included to further investigate how NTI164 works in the body.

DETAILED DESCRIPTION:
The FENRTT2 study will investigate the efficacy and safety of a full-spectrum medicinal cannabis plant extract with extremely low THC, NTI164, on Rett syndrome (RTT). This study will be a randomised, placebo-controlled, double-blind, crossover study spanning from 28 weeks up t0 52 weeks.

RTT is a devastating rare genetic condition affecting females and involves debilitating physical and intellectual symptoms, with inflammation often driving the progression of symptoms. NTI164 is a potently anti-inflammatory oil which has demonstrated efficacy in reducing symptoms in several paediatric neurological conditions, including RTT (Phase I/II), autism spectrum disorder (ASD), and paediatric acute-onset neuropsychicatric syndrome (PANS). A Phase I/II clinical trial of NTI164 in RTT (FENRTT1) showed NTI164 is safe in this population and significantly improved overall clinical severity of illness, as well as core RTT symptoms, including anxiety, mental alertness, communication skills, socialisation/eye contact, and attentiveness.

The FENRTT2 study will investigate NTI164 in a larger number of patients and will seek to demonstrate superiority over placebo in clinical outcomes in this cohort of patients. Multi-omic analyses on patient blood will also be included to further investigate the mechanism of action of NTI164, including transcriptomics, proteomics, phosphoproteomics, methylation, and cytokine analyses. Functional and clinical benefit will be measured using several validated, gold-standard assessment tools, rated by both clinicians and parents.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 4-25 years of age
2. Weight ≥12 kg
3. Classical/typical RTT as confirmed with a documented pathogenic variant in the MECP2 gene
4. At least 6 months post-regression at screening (i.e. no loss or degradation in ambulation, hand function, speech, non-verbal communication, or social skills within 6 months of screening)
5. Rett Syndrome Clinical Severity Scale rating of 10-36
6. Clinical Global Impression - Severity of Illness score ≥4
7. Stable pattern of seizures or has had no seizures within 8 weeks of screening, as determined by the participant's primary physician
8. Other patient medications must be stable (i.e. no dose adjustments) for at least 8 weeks prior to screening, including steroids, anti-inflammatories, anxiolytics etc

Exclusion Criteria:

1. Current clinically significant cardiovascular, endocrine (such as hypo- or hyperthyroidism, type 1 diabetes, or uncontrolled type 2 diabetes), renal, hepatic, respiratory, or gastrointestinal disease (such as coeliac disease or inflammatory bowel disease), or major surgery planned
2. Known history or symptoms of long QT syndrome
3. QTcF interval >450 milliseconds, history of risk factor for torsades de pointes or clinically significant QT prolongation deemed to increase risk
4. Currently receiving treatment with DAYBUE™ (Trofinetide)
5. Currently using other unregistered drugs for the treatment of Rett syndrome, such as Anavex®
6. Currently using or has used recreational or medicinal cannabis or cannabinoid-based medications, including Sativex® or Epidiolex®, within the 12 weeks prior to screening and is unwilling to abstain for the duration of the trial
7. A known or suspected hypersensitivity to cannabinoids or any of the excipients
8. Moderate-severe impairment in hepatic function at screening, defined as serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x upper limit of normal (ULN), or total bilirubin (TBL) > 2 x ULN. This criterion can only be confirmed once laboratory results are available, participants enrolled into the trial who are later found to meet this criterion will be screen-failed.
9. Participant is enrolled in another clinical trial within 14 days of screening or becomes enrolled in another clinical trial throughout the duration of this study
10. Infection and/or antibiotic use in the 2 weeks prior to screening (participants can be recruited following 2 weeks without infection and/or antibiotic use)

Ages: 4 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Rett Syndrome Behaviour Questionnaire (RSBQ) | Baseline, Week 12, and Week 28
  A validated, FDA-accepted 45-item caregiver-assessed tool to assess a variety of behavioural features impaired in RTT. The caregiver rates items as 0 = not true, 1 = somewhat true or sometimes true, or 2 = very true. Symptoms assessed include maladaptive behaviours, mood disruption, repetitive movements, fear/anxiety, breathing abnormalities, hand behaviours, and gross motor skills. A higher score indicates greater impairment/disease severity.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S) | Baseline, Week 12, and Week 28
  7-point scale rating a clinician's impression of disease severity at a given time point, a higher score indicates more severe illness.
Clinical Global Impression - Improvement (CGI-I) | Baseline, Week 12, and Week 28
  A clinician-rated tool to assess how much an individual's symptoms improve or worsen following an intervention on a 7-point scale. 1-3 = improvement, 4 = no change, 5-7 = worsening. It is anticipated the CGI-I score will be <4 following NTI164 treatment, indicating moderate-substantial improvement.
RTT-Domain- specific Concerns - Visual Analog Scale (RTT-DSC-VAS) | Baseline, Week 12, and Week 28
  An 8-point scale assessing areas of functional impairment (0 = normal function, 7 = most severe impairment).
Impact of Childhood Neurologic Disability scale + Quality of Life (ICND + QoL) | Baseline, Week 12, and Week 28
  Rates the effect of 4 health problems (inattentiveness, impulsivity, or mood; ability to think and remember; neurologic or physical limitations; epilepsy) on 11 aspects of the child and/or family's life (overall health, relationships with parents, relationships with siblings, relationship between your spouse/partner, relationships with child's friends/peers, social life - acceptability by others, social life - number of activities, school - academics, child's self-esteem, loss of original hopes for child/self, and family activities. A higher score indicates a lower level of disability. QoL component rates the QoL of the patient on a 6-point scale (1 = poor, 6 = excellent).
RTT-Caregiver Burden Inventory (RTT-CBI) | Baseline, Week 12, and Week 28
  Assesses 4 aspects of burden (physical, emotional, and social burden, and time dependence) on the primary caregiver of the patient. Subdomains include general caregiver tasks, emotional and social impact of caregiving, and financial burden. A higher score indicates greater impairment and caregiver burden.
EQ-5D-Y-5L | Baseline, Week 12, and Week 28
  A descriptive scale covering 5 dimensions of health (mobility, looking after myself, doing usual activities, having pain or discomfort, and feeling worried, sad, or unhappy). This version of the scale has 5 levels to each answer (5L) and is worded so as to be more child friendly (Y). A higher score indicates greater impairment/worse health status.
CSBS-DP-IT | Baseline, Week 12, and Week 28
  A caregiver rated scale often used as the first step in routine screening to determine if a developmental evaluation is needed. In the context of RTT, it can be used to assess functional communication. A higher score indicates a better communication ability.

OTHER OUTCOMES:
Research bloods - transcriptomics | Baseline, Week 12, Week 16, and Week 28
  To further clarify the mechanism of action of NTI164, both bulk and single-cell RNA sequencing will be performed on peripheral blood mononuclear cells (PBMCs) from patients at specified time points. This will provide additional information regarding which genes are being expressed in patients at either abnormally low or high levels compared to a non-RTT population, and the effects NTI164 has on gene expression. This workflow includes RNA extraction, depletion of ribosomal RNA via hybrid capture, library preparation, and sequencing. Cleaned sequence reads will then be aligned against the Homo sapiens genome (Build version hg38) and STAR aligner (v2.5.3a) will be used to map unique reads to the genomic sequences. This is exploratory so genes of interest cannot be identified in advance.
Research bloods - proteomics (and phosphoproteomics) | Baseline, Week 12, Week 16, Week 28
  To further clarify the mechanism of action of NTI164, proteomics and phosphoproteomics will be performed on peripheral blood mononuclear cells (PBMCs) from patients at specified time points. This will provide additional information regarding which proteins are being expressed at either abnormally low or high levels compared to a non-ASD population, as well as how extensively these proteins are phosphorylated compared to a non-ASD population, and the effects NTI164 has on protein expression and phosphorylation. Samples will be tagged using the TMTpro system and hydrophilic ion liquid chromatography fractionation performed. This is exploratory so proteins of interest cannot be identified in advance.
Research bloods - methylomics | Baseline, Week 12, Week 16, Week 28
  To further clarify the mechanism of action of NTI164, methylomics will be performed on whole blood from patients at specified time points. This will provide additional information on methylation patterns (e.g. addition of a methyl group to histones or DNA) in patients compared to non-patients, and how NTI164 effects this type of epigenetic modification and how genes of interest may be regulated. This is exploratory so patterns of interest cannot be identified in advance. Genome-wide methylation will be assessed using the Illumina MethylationEPIC v2.0 BeadChip (or the latest version if a new version is available to the study team at the time of analysis).
Research bloods - cytokine assay | Baseline, Week 12, Week 16, Week 28
  To further clarify the mechanism of action of NTI164, a cytokine assay investigating a panel of inflammatory markers will be performed on plasma from patients at specified time points. The cytokine assay will likely be the LEGENDplex Human Neuroinflammation Panel 1 (13 plex). Cytokines investigated with this panel include VILIP-1, CCL2, sTREM-2, b-NGF, TGF-b1, TNF-a, IL-6, s-TREM-1, sRAGE, CX3CL1, VEGF, BDNF, and IL-18.

CONTACTS AND LOCATIONS:
Locations (1):
- Monash Health, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No